CLINICAL TRIAL: NCT06472934
Title: Impact of Beta-blocker Administration on Outcome Among Patients Undergoing Transcatheter Aortic Valve Replacement B-TAVR
Brief Title: Impact of Beta-blocker on Outcome Among Patients Undergoing Transcatheter Aortic Valve Replacement (B-TAVR)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00728; kt23Nestelberger2
Record Dates: First submitted 2024-06-13; First posted 2024-06-25 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Aortic Stenosis
Keywords: Transcatheter Aortic Valve Replacement; Beta-blockers
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pausing group (Experimental): Subjects in the pausing group will stop their B-blocker medication 72h before the scheduled transcatheter aortic valve replacement (TAVR) procedure. Post-procedural B-blocker therapy will be resumed 72h after the procedure using the same type and dosage as prescribed before.
  Interventions: Other: Transcatheter aortic valve replacement in the absence of B-blocker treatment
- Control group (Other): Subjects in the control group will keep their B-blocker medication in their prescribed dose during the scheduled TAVR procedure.
  Interventions: Other: Transcatheter aortic valve replacement

INTERVENTIONS:
Other: Transcatheter aortic valve replacement in the absence of B-blocker treatment — Transcatheter aortic valve replacement (TAVR) is performed in patients that temporarily pause B-blocker treatment.
  Arms: Pausing group
Other: Transcatheter aortic valve replacement — Transcatheter aortic valve replacement (TAVR) is performed in patients that do not temporarily pause B-blocker treatment.
  Arms: Control group

SUMMARY:
This is a multi-centric, open-label, randomized trial to evaluate the safety and efficacy of temporary discontinuation of beta-blocker treatment in patients undergoing transcatheter aortic valve replacement.

DETAILED DESCRIPTION:
Aortic stenosis (AS) is a common heart valve problem in older adults, affecting about 5% of people over 65. It leads to symptoms like fainting, chest pain, difficulty breathing, and heart failure, which can increase the risk of serious health issues and death.

Transcatheter Aortic Valve Replacement (TAVR) is a well-established treatment for severe AS, especially for patients who are at high risk for traditional open-heart surgery. TAVR is becoming more common and is now being used in younger and lower-risk patients due to its favorable outcomes.

Many people with severe AS also have other heart conditions, and beta-blockers (B-blockers) are commonly used to manage these issues. B-blockers help treat heart failure, irregular heartbeats, high blood pressure, and coronary artery disease. About 34% to 51% of AS patients use B-blockers, but these medications can also cause side effects like slow heart rate and low blood pressure.

The need for a permanent pacemaker is the most common complication after TAVR, occuring in 9% to 26% of patients. This is because TAVR can affect the heart's electrical system. B-blockers might increase the risk of needing a pacemaker because they can further slow down the heart's electrical signals.

To reduce this risk, doctors sometimes stop B-blockers around the time of TAVR. However, this practice lacks support from clinical trials or guidelines, and stopping B-blockers can increase the risk of fast heartbeats and chest pain.

This aim of the clinical trial is to study the impact of B-blocker administration among patients undergoing TAVR. The trial will assess the safety of B-blocker discontinuation (primary endpoint) and by determining the incidence of permanent pacemaker implantation after TAVR (secondary endpoint).

The results of the trial will provide important insights into the optimal management of B-blockers in patients undergoing TAVR, potentially improving patient outcomes and guiding clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent must be signed by the subject prior to any study intervention.
* Adult patients (> 18 years) with severe symptomatic aortic stenosis eligible and scheduled for elective TAVR and are able to give consentand are able to give consent
* Indication for B-blocker therapy with a prior treatment duration of at least 1 month before inclusion.

Exclusion Criteria:

* Emergency or urgent indication for TAVR.
* Hemodynamically unstable patients receiving inotropic medication.
* Prior permanent pacemaker implantation.
* Existing indication for pacemaker implantation.
* Hemodynamic relevant left ventricular outflow tract obstruction.
* Prior intolerance of B-blocker medication.
* Life expectancy < 1 year.
* Known or suspected non-compliance, drug, or alcohol abuse.
* Inability to give consent, or follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Being in a dependent relationship with the trial site
* Participation in another study with investigational drug within the 30 days preceding and during the present study.
* Previous enrolment into the current study.
* Pregnancy or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | At 30 days
  To analyse the safety of B-blocker discontinuation, the all-cause mortality, as part of a composite endpoint, is assessed within 30 days after transcatheter aortic valve replacement (TAVR).
Re-hospitalization due to heart failure | At 30 days
  To analyse the safety of B-blocker discontinuation, the incidence of re-hospitalization due to heart failure, as part of a composite endpoint, is assessed within 30 days after TAVR.
  Re-hospitalization due to heart failure is defined as an admission occurring after the index hospitalization or study enrollment, where new or worsening heart failure is the primary reason for a hospital stay exceeding 24 hours. This determination is based on symptoms and signs of heart failure, confirmed by diagnostic tests, and requires treatment with intravenous or mechanical heart failure therapies. This includes both primary (cardiac-related) and secondary (non-cardiac-related) causes.
Stroke Rate | At 30 days
  To analyse the safety of B-blocker discontinuation, the incidence of stroke, as part of a composite endpoint, is assessed within 30 days after TAVR.
Severe arrhythmia requiring treatment | At 30 days
  To analyse the safety of B-blocker discontinuation, the incidence of severe arrhythmia that requires treatment, as part of a composite endpoint, is assessed within 30 days after TAVR.
  Severe arrhythmia requiring treatment are e.g. new onset atrial fibrillation/flutter, ventricular tachycardia/ventricular fibrillation, new atrioventricular block (AB, first-, second- or third-degree), new left bundle branch block, new right bundle branch block, new severe bradycardia or tachycardia (<40bpm or >120bpm).

SECONDARY OUTCOMES:
Permanent pacemaker implantation Rate | At 30 days and 1 year
  To analyse the efficacy of B-blocker discontinuation, the incidence of permanent pacemaker implantation is assessed within 30 days and 1 year after TAVR.
Stroke Rate | At 30 days and 1 year
  The incidence of stroke is assessed within 30 days and 1 year after TAVR.
All-cause mortality | At 30 days and 1 year
  The all-cause mortality is assessed within 30 days and 1 year after TAVR.
Cardiovascular mortality | At 30 days and 1 year
  The cardiovascular mortality is assessed within 30 days and 1 year after TAVR. It is defined as either:
  * Related to heart failure, cardiogenic shock, bioprosthetic valve dysfunction, myocardial infarction, stroke, thromboembolism, bleeding, tamponade, vascular complication, arrhythmia or conduction system disturbances, cardiovascular infection (e.g. mediastinitis, endocarditis),or other clear cardiovascular cause
  * Intraprocedural death
  * Sudden death
  * Death of unknown cause
Re-hospitalization due to heart failure | At 30 days and 1 year
  The incidence of re-hospitalization due to heart failure, as part of a composite endpoint, is assessed within 30 days and 1 year after TAVR.
  Re-hospitalization due to heart failure is defined as an admission occurring after the index hospitalization or study enrollment, where new or worsening heart failure is the primary reason for a hospital stay exceeding 24 hours. This determination is based on symptoms and signs of heart failure, confirmed by diagnostic tests, and requires treatment with intravenous or mechanical heart failure therapies. This includes both primary (cardiac-related) and secondary (non-cardiac-related) causes.
Severe arrhythmia requiring treatment | At 30 days and 1 year
  The incidence of severe arrhythmia that requires treatment, as part of a composite endpoint, is assessed within 30 days and 1 year after TAVR.
  Severe arrhythmia requiring treatment are e.g. new onset atrial fibrillation/flutter, ventricular tachycardia/ventricular fibrillation, new atrioventricular block (AB, first-, second- or third-degree), new left bundle branch block, new right bundle branch block, new severe bradycardia or tachycardia (<40bpm or >120bpm).

OTHER OUTCOMES:
Health economic assessment | At 30 days and 1 year
  An assessment of the impact on health economic is performed, which includes information regarding the length of intensive care unit stay, length of hospital stay, rate of pacemaker implantation, and results of the Kansas City Cardiomyopathy quality of life Questionnaire (KCCQ-12) which ranges from 0 to 100 with higher scores indicating better health status and quality of life, while lower scores suggest more severe symptoms and poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Nestelberger, PD Dr., Principal Investigator — University Hospital Basel, Department of Cardiology & Cardiovascular Research Institute Basel (CRIB)
Locations (11):
- Austria (2):
  - Medical University of Graz, Graz
  - University Hospital Salzburg, Salzburg
- Germany (5):
  - University Medical Center Freiburg, Bad Krozingen
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Herz- und Diabeteszentrum NRW Universitätsklinik, Bad Oeynhausen
  - Universitätsklinikum Giessen und Marburg GmbH, Giessen
  - Universitätsklinikum Schleswig-Holstein AöR, Kiel
- Switzerland (4):
  - University Hospital Basel, Basel
  - Inselspital, Bern University Hospital, Bern
  - Geneva University Hospitals, Geneva
  - University Hospital of Zürich, Zurich